CLINICAL TRIAL: NCT04066400
Title: Role of a Wheat-based Diet in NASH (NASH-ATI)
Brief Title: Role of a Wheat Containing Diet on Non-alcoholic Steatohepatitis
Acronym: NASH-ATI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johannes Gutenberg University Mainz (Other)
Collaborators: Goethe University (Other)
Responsible Party: Principal Investigator, Jörn M. Schattenberg, Director Metabolic Liver Disease Program, Johannes Gutenberg University Mainz
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2018-13078
Record Dates: First submitted 2019-08-17; First posted 2019-08-26 (Actual); Last update posted 2023-12-28 (Actual); Status verified 2023-12

CONDITIONS: NASH - Nonalcoholic Steatohepatitis; Diabetes Mellitus, Type 2; Hyperlipidemias
Keywords: hepatic inflammation
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease; Diabetes Mellitus, Type 2; Hyperlipidemias

STUDY DESIGN:
Intervention Model Description: prospective, randomized, controlled, bicentric pilot study
Who Masked: Outcomes Assessor
Masking Description: randomization
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- wheat-based diet (Placebo Comparator): The patients continue a wheat-based diet aiming at a reduction in bodyweight.
  Interventions: Other: Nutritional Intervention
- ATI reduced diet (Experimental): Patients are counselled to reduce dietary gluten uptake.
  Interventions: Other: Nutritional Intervention

INTERVENTIONS:
Other: Nutritional Intervention — Dietary Counselling

SUMMARY:
Effects of Wheat-based diet vs. ATI-free diet on NASH

DETAILED DESCRIPTION:
40 patients with the diagnosis of a non-alcoholic- steatohepatitis (NASH) will be recruited at the University Hospitals of Mainz and Frankfurt. Patients are assessed with regards to their diet using standardized questionnaire and nutritionists.

Patients will be randomized into two parallel groups. The first group will continue a wheat-based Nutrition, while the second Group will receive dietary counselling to achieve an ATI-free nutrition, trying to reduce the daily ATI consumption.

The clinical trial will run over 16 weeks including 4 visits at the study center. Study visits include physical examinations, blood-based parameters, cytokines and urine samples, as well for the analysis of the intestinal microbiome by using stool samples. In addition the patients have to complete dietary and health-related quality of life (HRQL) questionnaires. Visits are planned at baseline, W4, W8 and W16.

ELIGIBILITY:
Inclusion Criteria:

* histologically proven NASH in the past 36 months with increased ALT: males: >60, females: >42 U/ml
* no body weight modification about >10% in the past 24 weeks
* no new drugs treating parts of the metabolic syndrome in the past 12 weeks
* for patients with Diabetes: HbA1c value <8,6%
* the ability to understand the aim and the possible individual consequences of this Trial
* signed and dated consent before the Trial starts

Exclusion Criteria:

* unstable coronary heart disease, stroke in the past 6 months
* different liver diseases
* proceeded fibrosis (Fibroscan >9,6 kPA) or histological cirrhosis
* hepatocellular carcinoma or not curative treated carcinomas
* alcohol consumption >10g/day (females), >20g/day (males)
* gravidity
* drugs causing secondary NASH (e.g. Tamoxifen, corticosteroids)
* immunological or inflammatory diseases (e.g. systemic Lupus erythematodes)
* warfarin therapy
* implementation of another Special diet

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2018-10-01 (Actual); Primary Completion 2022-01-01 (Actual); Study Completion 2023-12-27 (Actual)

PRIMARY OUTCOMES:
Effect of ATI-free Nutrition on hepatic inflammation | 16 weeks
  Reduction of Alanine-Aminotransferase (ALT; U/ml) compared to baseline

SECONDARY OUTCOMES:
Quality of Life using the chronic liver disease questionnaire (CLDQ) | 16 weeks
  The CLDQ is a validated patient-reported outcome measure

CONTACTS AND LOCATIONS:
Locations (2):
- Germany (2):
  - Universität Frankfurt, Frankfurt
  - University Medical Center Mainz, Mainz

REFERENCES:
- [Derived] Armandi A, Bespaljko H, Mang A, Huber Y, Michel M, Labenz C, Galle PR, Neerukonda M, Bugianesi E, Schuppan D, Schattenberg JM. Short-term reduction of dietary gluten improves metabolic-dysfunction associated steatotic liver disease: A randomised, controlled proof-of-concept study. Aliment Pharmacol Ther. 2024 May;59(10):1212-1222. doi: 10.1111/apt.17941. Epub 2024 Mar 11. PMID 38462919